CLINICAL TRIAL: NCT04477408
Title: Effect of Plantar Sensory Exercises on Balance and Fall Risk in Nursing Home Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, muyesser cavlak, Chief Researcher, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulMUH - 2
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2020-07

CONDITIONS: Balance; Distorted; Plantar; Falling; Elderly; Sensitivity
Keywords: plantar sensation, balance, fall, elderly
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: self controlled prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plantar exercise group (Other): plantar sensitive exercises
  Plantar sensitive exercises:
  30 minutes / 3 days per week / 8 weeks Walking on different 4 different textured floors and hot floor (15 minute) Trying to recognize small objects with the soles of the feet (5min) Seated work with barbed ball and balance pad (5min) Massage to the sole of the foot with different textured fabrics (5min)
  Interventions: Other: plantar sensory exercise group

INTERVENTIONS:
Other: plantar sensory exercise group — plantar sensitive exercises
  Plantar sensitive exercises:
  30 minutes / 3 days per week / 8 weeks Walking on different 4 different textured floors and hot floor (15 minute) Trying to recognize small objects with the soles of the feet (5min) Seated work with barbed ball and balance pad (5min) Massage to the sole of the foot with different textured fabrics (5min)

SUMMARY:
The most important cause of mortality and morbidity with the geriatric population is loss of balance and the consequent falls, which is seen very often. The goal of our study is to examine the effects of plantar sensation education-based exercises on balance and falls.Materials and methods: 16 healthy, voluntary nursing home residents with the average age 77.50±5.5. Individuals had plantar sensory exercises 40 min sessions for 3 days/week during eight weeks. The study was planned as a self-controlled prospective study. Functional balance was evaluated using Berg Balance Scale, dynamic balance was evaluated using 30 Second Chair Stand Test, static balance and fall risk were assessed using Biodex Balance System.

DETAILED DESCRIPTION:
The study was run in Istanbul Provincial Directorate of Social Services Istanbul Prof. Dr. Fahrettin Kerim-Nilüfer Gökay Nursing Home Elderly Care and Rehabilitation Center in March-June 2019. This study was designed as a self-controlled prospective non-randomized study.

Written informed consent was obtained from all participants. The necessary ethical approval for the study was taken from the Medipol University Non-Interventional Clinical Research Ethics Comittee This study was planned to be run with 20 healthy nursing home residents. The criteria of being included in the study were: being above 70 years of age, scoring at least 22 points on the Mini Mental Test, not being bound to a wheelchair, being able to walk 20 meters independently, and that the sensation of the foot sole is at least on the decreased protective level compare to Semmes Weinstein Monofilamnet test. The individuals with serious loss of eyesight, mental retardation, a schizophrenic background, having walking disorder, inconvenient in walking were not included in the study.

16 healthy aged individuals with the average age of 77.50±5.5 participated in our study. 2 of the first 20 participants left the study due to health problems and 2 other participants left due to personal reasons which they did not want to declare (Figure 1).

A homogeneous control group could not be created due to aging, so a control group was created with the same participants. The first evaluations of our study were made within two days. After the evaluation process, 4 weeks waiting period was given. At the end of this period, second measurements were made for two days. Plantar sensory based exercises program lasting 8 weeks was applied after the second measurements were taken. Post-treatment measurements were made for two days after the treatment ended. Measurements were made with MC and the physiotherapist working in the nursing home.

ELIGIBILITY:
Inclusion Criteria:

* Being above 70 years of age
* Scoring at least 22 points on the Mini Mental Test
* Not being bound to a wheelchair
* Being able to walk 20 meters independently
* That the sensation of the foot sole is at least on the decreased protective level compare to Semmes Weinstein Monofilamnet test.

Exclusion Criteria:

* Serious loss of eyesight
* Mental retardation
* A schizophrenic background
* Having walking disorder
* Inconvenient in walking

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Biodex Balance System - Static Balance | 0 week
  The device calculates a score of stability or loss of balance in the anteroposterior and mediolateral direction. It also calculates an average stability index by taking the average of these two scores. The general balance index score was used which was obtained according to the protocol in the guide manual of the device. The measurement of static balance was repeated 3 times on the 8th level mode with a test duration of 30 seconds, with 15 seconds of rest periods and the best result was taken into evaluation. A high score indicates that the loss of postural control and balance is high.
Biodex Balance System - Static Balance | 4 week
  The device calculates a score of stability or loss of balance in the anteroposterior and mediolateral direction. It also calculates an average stability index by taking the average of these two scores. The general balance index score was used which was obtained according to the protocol in the guide manual of the device. The measurement of static balance was repeated 3 times on the 8th level mode with a test duration of 30 seconds, with 15 seconds of rest periods and the best result was taken into evaluation. A high score indicates that the loss of postural control and balance is high.
Biodex Balance System - Static Balance | 12 week
  The device calculates a score of stability or loss of balance in the anteroposterior and mediolateral direction. It also calculates an average stability index by taking the average of these two scores. The general balance index score was used which was obtained according to the protocol in the guide manual of the device. The measurement of static balance was repeated 3 times on the 8th level mode with a test duration of 30 seconds, with 15 seconds of rest periods and the best result was taken into evaluation. A high score indicates that the loss of postural control and balance is high.
Biodex Balance System - Fall Risk | 0 week
  For evaluate to fall risk the device was used as stated in the guide manual. The test was run gradually by moving from an unstable surface to a stable surface for 20 seconds in three sets. Between each set, the participants rested for 10 seconds. A high score indicates that the fall risk is high.
Biodex Balance System - Fall Risk | 4 week
  For evaluate to fall risk the device was used as stated in the guide manual. The test was run gradually by moving from an unstable surface to a stable surface for 20 seconds in three sets. Between each set, the participants rested for 10 seconds. A high score indicates that the fall risk is high.
Biodex Balance System - Fall Risk | 12 week
  For evaluate to fall risk the device was used as stated in the guide manual. The test was run gradually by moving from an unstable surface to a stable surface for 20 seconds in three sets. Between each set, the participants rested for 10 seconds. A high score indicates that the fall risk is high.

SECONDARY OUTCOMES:
Berg Balance Scale | 0 week
  This test evaluates the individuals' ability to maintain their balance during functional activity. Berg Balance Scale is run with 14 different activities. A score between 0-20 shows high risk, a score between 21-40 shows medium risk and a score between 41-64 shows low risk
Berg Balance Scale | 4 week
  This test evaluates the individuals' ability to maintain their balance during functional activity. Berg Balance Scale is run with 14 different activities. A score between 0-20 shows high risk, a score between 21-40 shows medium risk and a score between 41-64 shows low risk
Berg Balance Scale | 12 week
  This test evaluates the individuals' ability to maintain their balance during functional activity. Berg Balance Scale is run with 14 different activities. A score between 0-20 shows high risk, a score between 21-40 shows medium risk and a score between 41-64 shows low risk
30 Second Chair Stand Test | 0 week
  30 Second Chair Stand Test evaluates an individuals' dynamic balance with their activity of sitting and standing up. It is performed by asking the participant to constantly sit down and stand up from a chair within 30 seconds and noting how many times they do it.
30 Second Chair Stand Test | 4 week
  30 Second Chair Stand Test evaluates an individuals' dynamic balance with their activity of sitting and standing up. It is performed by asking the participant to constantly sit down and stand up from a chair within 30 seconds and noting how many times they do it.
30 Second Chair Stand Test | 12 week
  30 Second Chair Stand Test evaluates an individuals' dynamic balance with their activity of sitting and standing up. It is performed by asking the participant to constantly sit down and stand up from a chair within 30 seconds and noting how many times they do it.

CONTACTS AND LOCATIONS:
Overall Officials: Müyesser Cavlak, Study Chair — İstanbul Medipol University; Candan Algun, Prof, Study Director — İstanbul Medipol University
Locations (1):
- İstanbul Medipol University, Istanbul, Kavacık, Turkey (Türkiye)